CLINICAL TRIAL: NCT04915911
Title: A Multi-center, Cross-sectional Observational Study on Nutritional Status and Body Composition of Adult Patients With Crohn's Disease
Brief Title: Nutritional Status and Body Composition of Adult Patients With Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1109
Record Dates: First submitted 2021-04-11; First posted 2021-06-07 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with Crohn's disease: multi-center cross-sectional study
  Interventions: Other: cross-sectional study

INTERVENTIONS:
Other: cross-sectional study — cross-sectional study

SUMMARY:
Patients with Crohn's disease generally have nutritional risks and malnutrition. The investigators will conduct a multicenter cross-sectional study to discover nutritional status and body composition of Chinese adult patients with CD.

DETAILED DESCRIPTION:
Several studies have found that the body composition of CD patients is related to disease and therapies. Due to lack of a prospective multicenter cross-sectional observational study on the nutritional status and body composition of adult patients with CD in China. Evaluating the nutritional status and body composition of these patients can help formulate individualized nutritional support strategies for adult CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* diagnosis of CD;
* Admission time <48 hours;
* Subject has voluntarily signed and dated an informed consent form.

Exclusion Criteria:

* Emergency surgery for intestinal fistula or abdominal abscess;
* Unstable vital signs or unstable hemodynamics;
* Pregnant or lactating women;
* Admission to hospital due to other critical illnesses (such as tumor, HIV, severe infections requiring ventilator or CRRT treatment);
* Dying patients whose life expectancy does not exceed 24 hours;
* Severe liver insufficiency (liver function score 11-15 or total bilirubin> 3mg/dL or tissue biopsy diagnosed as liver cirrhosis, hepatic encephalopathy, portal hypertension with history of gastrointestinal hemorrhage, etc.);
* Severe renal insufficiency (creatinine value is 2 times higher than the upper limit of normal);
* Severe metabolic diseases (such as metabolic syndrome, hyperthyroidism, etc.);
* Patients whose burn area exceeds 20% of the body surface area;
* Immunodeficiency, autoimmune disease, or receiving immunosuppressive treatment for diseases other than CD (such as organ transplantation, etc.);
* Those who are not suitable for body composition analysis
* Patients who have been selected for other clinical studies or have been selected for this study;
* Subjects are unwilling to participate in this study or refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult patients with Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal mass index | Within 48 hours of admission to hospital
  Bioelectrical impedance analysis

SECONDARY OUTCOMES:
Body composition | Within 48 hours of admission to hospital
  Especially body fat mass by bioelectrical impedance analysis
Nutritional risk screening | Within 48 hours of admission to hospital
  Detect the presence of undernutrition and the risk of developing undernutrition by Risk Screening 2002 (NRS-2002), when score≥3, the patient is nutritionally at-risk
Nutritional assessment | Within 48 hours of admission to hospital
  Detect malnourished individuals by the Subjective Global Assessment (SGA) , where A is well nourished and C is severely malnourished
Grip strength | Within 48 hours of admission to hospital
  Hand grip strength test

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China